CLINICAL TRIAL: NCT05213689
Title: Kuwawezesha Vijana (Empowering Youth): An HIV Self-Testing and Comic Intervention With Refugee Adolescents and Youth in a Refugee Settlement in Northern Uganda
Brief Title: HIV Self-Testing and Comic Intervention With Refugee Adolescents and Youth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Carmen Logie, MSW, PhD, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: bidibidi_viiv
Record Dates: First submitted 2022-01-27; First posted 2022-01-28 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: HIV/AIDS; HIV Infections; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Behavior

STUDY DESIGN:
Intervention Model Description: This cluster-randomized controlled trial (RCT) will evaluate the effectiveness of HIVST delivery approaches on HIV testing uptake among refugee youth in the Bidi Bidi Refugee Settlement. Participants from two villages within each of the two zones (i.e., four geographically different areas) will be randomized together to one of 4 study arms: Arm 1-HIVST, Arm 2- HIVST+ educational comic book, Arm 3-educational comic book, and Arm 4 - standard of care(control). Data collectors will administer tablet-based surveys (baseline and at 3 months).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIV self-testing + educational comic book (Experimental): At the first visit participants will receive a HIVST kit and a detailed description of how to use the HIVST kits, pictorial and written guide for HIVST kits, in addition to contact information for confirmatory testing and linkage to care at local clinics. Participants will also receive an educational comic book focused on HIV testing information and decision making that was developed with qualitative data collected from an earlier study phase. PNs will meet with small groups of participants to read through and discuss the comic book together.
  Interventions: Behavioral: Educational comic book; Diagnostic Test: HIV Self-testing
- HIV self-testing (Active Comparator): At the first visit participants will receive a HIVST kit and a detailed description of how to use the HIVST kits, pictorial and written guide for HIVST kits, in addition to contact information for confirmatory testing and linkage to care at local clinics.
  Interventions: Diagnostic Test: HIV Self-testing
- Educational comic book (Active Comparator): Participants will receive an educational comic book focused on HIV testing information and decision making that was developed with qualitative data collected from an earlier study phase. PNs will meet with small groups of participants to read through and discuss the comic book together.
  Interventions: Behavioral: Educational comic book
- Standard of Care (No Intervention): PNs will provide information about HIV testing, care and support services at local clinics.

INTERVENTIONS:
Behavioral: Educational comic book — An educational comic book was developed with qualitative data collected from an earlier study phase involving focus groups with youth from Bidi Bidi. The comic book is focused on HIV testing information and decision making as it follows the story of youth in Bidi Bidi who are seeking out HIV testing. Each youth in the appropriate arm with receive a copy of the comic book and together with 5-10 other youth will meet with a PN to read through and discuss the comic book. The comic will also include blank pages so that the youth can participate in the dialogue of the comic book. The comic will be available in English, Bari and Juba Arabic.
  Arms: Educational comic book; HIV self-testing + educational comic book
Diagnostic Test: HIV Self-testing — Participants will receive HIVST kits so that they can perform their HIV testing.
  Arms: HIV self-testing; HIV self-testing + educational comic book

SUMMARY:
HIV is the leading cause of death for adolescents and young people (AYP) in sub-SaharanAfrica (SSA). Uganda hosts 1.4 million refugees/displaced persons and the Bidi Bidi refugee camp in Northern Uganda is the second-largest refugee settlement in the world and the largest in Africa. There are reports of high sexual and gender-based violence (SGBV) among refugees during the journey from South Sudan to Uganda and in the refugee settlements, yet low rates of HIV testing and access to HIV prevention services, particularly tailored for gender, age, and the refugee settlement context. This study aims to develop, implement and evaluate an oral HIV-self testing (HIVST) intervention with displaced/refugee AYP aged16- 24 in Bidi Bidi. HIVST is acceptable and properly used with AYP in other SSA regions, yet there are knowledge gaps regarding the best way to link HIVST to HIV care. This study aims to explore how user-developed educational comic books can improve linkage to care with HIVST. This trial focuses on implementing a randomized trial with displaced/refugee AYP aged 16-24 living in Bidi Bidi (Arm1: HIVST; Arm 2: HIVST + comic book; Arm 3: comic book; Arm 4: standard of care). The study will assess changes in HIV testing practices, HIV status knowledge, and linkage to HIV prevention and care between the 4 arms.

DETAILED DESCRIPTION:
The proposed study will take place in Bidi Bidi Refugee Settlement within Yumbe district in northwestern Uganda, hosting over 200,000 refugees.This research will be conducted in Zone 3 and 5 in Bidi Bidi. The proposed intervention involves a randomized controlled trial (RCT) to evaluate the effectiveness of HIVST delivery approaches on HIV testing uptake among refugee youth aged 16-24 in Bidi Bidi. Participants will be cluster-randomized in one of four study arms (Arm 1: HIVST; Arm 2: HIVST + comic book; Arm 3: comic book; Arm 4: standard of care). Participants from specific villages within two Bidi Bidi zones will be randomized to an arm together.

HIVST Interventions (Arm 1 and 2): At the first visit study participants are provided with a HIVST kit (Oraquick: approved and used in Uganda by the Ministry of Health) that is an oral swab test stick and tube solutions, and a written detailed step by step description of how to correctly use the HIVST kits, pictorial and written guide for HIVST kits, information on HIV and testing, referral cards with addresses and phone numbers to local clinics for confirmatory testing. The cards will also have a peer navigator (PN)'s phone numbers for participants to call or text message (SMS) if they need additional information on how to use the kits, or support to go to confirmatory tests at the clinics. Instructions for the kits are in English, Bari and Juba Arabic and reflect the context of the rural displaced adolescent and young people. The Research Coordinator and PN team will rotate being on-call to respond to any issues by text and will offer to phone or text support the participant and offer to make an appointment to see them and/or support them to attend a collaborating clinic for further support.

Educational comic book (Arm 2 and 3): Participants will receive an educational comic book focused on HIV testing information and decision making that was developed with qualitative data collected from an earlier study phase. PNs will meet with small groups of participants to read through and discuss the comic book together.

Standard of Care: PNs will provide information about HIV testing, care and support services at local clinics.

Participant retention: Community collaborators will facilitate recruitment and retention; PNs will use multiple study reminder strategies (e.g. social media, texts) to maintain engagement, and we will utilize existing outreach and services by Uganda Refugee and Disaster Management Council (URDMC).

Research Team Training: This research involves collaborations with local clinics and URDMC in Bidi Bidi. Clinic staff will provide technical assistance for HIVST and train PN and the research team in: a) using HIV rapid test kits (Alere Determine HIV-1/2); b) using OraQuick, a rapid oralHIVST used in Uganda; c) pre/post HIV test counselling; and d) linkages to confirmatory testing and HIV care.

Linkage to testing and care: Participants across all study arms will meet with PN at two timepoints (t0: baseline, t1: 3 months) to complete surveys. Each participant will have a study identification (ID) number printed on 'movie coupons'; they can bring these coupons to clinics for HIV testing, confirmatory testing, linkage to HIV care, sexual and reproductive health services.The survey ID will be linked to resources accessed. Persons who test positive will be linked with local support groups and services, which have been identified and will the linkage be facilitated by local collaborators URDMC.

ELIGIBILITY:
Inclusion Criteria:

* living in one of the selected villages in Zone 3 & 4 Annex in the Bidi Bidi Refugee Settlement
* identify as a refugee/displaced person or have refugee parents
* aged 16-24 years

Exclusion Criteria:

* do not identify as a refugee or do not have refugee parents
* do not live in the selected villages in Zone 3 & 4 Annex

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Changes in HIV testing frequency | Time 1 (month 0), Time 2 (month 3)
  To assess changes in past 3 month HIV testing frequencies, participants are asked to self-report when their last HIV test was and where their last HIV test was (if they used the HIVST, clinic, or point-of-care testing).
HIV status knowledge | Time 2 (month 3)
  At the final 3-month visit, a clinician supported by trained peer navigators will offer all participants a completely voluntary rapid point-of-care HIV test (Alere Determine HIV-½) to measure HIV status knowledge. HIV status knowledge will be assessed as correct for participants that agree to take the rapid test and correctly report their HIV status before receiving the result.

SECONDARY OUTCOMES:
Linkage to confirmatory HIV testing | Time 2 (month 3)
  Interviewer will ask HIVST arms if they used their HIVST kit, for those who did, we will ask result. For those reporting a positive result we will ask if/where they received confirmatory testing. Participants can also submit coupons at collaborating health clinics with coupons with their study ID# for confirmatory tests that can be linked to study.
Change in HIV-related stigma | Time 1 (month 0), Time 2 (month 3)
  Attitudes and beliefs towards HIV will be assessed using Steward et al., (2008) HIV-related stigma scale including vicarious and felt-normative HIV stigma dimensions.
Change in HIV knowledge | Time 1 (month 0), Time 2 (month 3)
  HIV knowledge will be assessed using 18-item brief HIV knowledge questionnaire by Carey & Schroder, 2002.
Change in access to other sexual and reproductive health services | Time 1 (month 0), Time 2 (month 3)
  Interviewer will ask all participants to self-report their use of condoms (at time of last sex, % of times during sex in past 1 month), use of contraception [or partner's use for men] (current use [yes/no], type). Participants can also submit coupons at collaborating health clinics with coupons with their study ID# for SRH services that can be linked to study.
Linkage to HIV care | Time 2 (month 3)
  Participants who seroconvert in the study will be asked if they received HIV care, including ART and counseling, since receiving an HIV-positive diagnosis.
HIV self-test kit use | One month after Time 2
  In order to understand the use of HIV self-test kits and to reduce social desirability bias, one month after Time 2 the participants in arm 1 and arm 2 will be asked if they have unused test kits. They will be informed this information is just to guide future trials.
Safer sex efficacy | Time 1 (month 0), Time 2 (month 3)
  Measured using the Condom Use Self-Efficacy Scale (Shaweno et al., & Brafford et al.)
Condom use | Time 1 (month 0), Time 2 (month 3)
  Measured using questions asking about condom use at last sex; condom use at sex every time in last 3 months [dichotomous: yes/no]
Adolescent sexual and reproductive health stigma | Time 1 (month 0), Time 2 (month 3)
  Assessed with the Ugandan Adolescent Sexual and Reproductive Health (SRH) Stigma scale (Logie et al. 2019) adapted from Hall et al.'s Adolescent SRH Stigma scale
Sexual relationship power | Time 1 (month 0), Time 2 (month 3)
  Measured using Relationship Control Sub-Scale from the Sexual & Relationship Power Scale (Pulerwitz et al.)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Logie, PhD, Principal Investigator — University of Toronto
Locations (1):
- Factor-Inwentash Faculty of Social Work, University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Background] Steward WT, Herek GM, Ramakrishna J, Bharat S, Chandy S, Wrubel J, Ekstrand ML. HIV-related stigma: adapting a theoretical framework for use in India. Soc Sci Med. 2008 Oct;67(8):1225-35. doi: 10.1016/j.socscimed.2008.05.032. Epub 2008 Jul 1. PMID 18599171
- [Background] Carey MP, Schroder KE. Development and psychometric evaluation of the brief HIV Knowledge Questionnaire. AIDS Educ Prev. 2002 Apr;14(2):172-82. doi: 10.1521/aeap.14.2.172.23902. PMID 12000234
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Shaweno D, Tekletsadik E. Validation of the condom use self-efficacy scale in Ethiopia. BMC Int Health Hum Rights. 2013 Apr 23;13:22. doi: 10.1186/1472-698X-13-22. PMID 23617404
- [Background] Brafford LJ, Beck KH. Development and validation of a condom self-efficacy scale for college students. J Am Coll Health. 1991 Mar;39(5):219-25. doi: 10.1080/07448481.1991.9936238. PMID 1783705
- [Background] Pulerwitz J, Gortmaker SL, Dejong W. Measuring Sexual Relationship Power in HIV/STD Research. Sex Roles. 2000;42:637-60.
- [Background] Hall KS, Manu A, Morhe E, Harris LH, Loll D, Ela E, Kolenic G, Dozier JL, Challa S, Zochowski MK, Boakye A, Adanu R, Dalton VK. Development and Validation of a Scale to Measure Adolescent Sexual and Reproductive Health Stigma: Results From Young Women in Ghana. J Sex Res. 2018 Jan;55(1):60-72. doi: 10.1080/00224499.2017.1292493. Epub 2017 Mar 7. PMID 28266874
- [Background] Logie CH, Okumu M, Mwima SP, Kyambadde P, Hakiza R, Kibathi IP, Kironde E, Musinguzi J, Kipenda CU. Exploring associations between adolescent sexual and reproductive health stigma and HIV testing awareness and uptake among urban refugee and displaced youth in Kampala, Uganda. Sex Reprod Health Matters. 2019 Dec;27(3):86-106. doi: 10.1080/26410397.2019.1695380. PMID 31880507
- [Derived] Logie CH, Okumu M, Loutet MG, Coelho M, Berry I, Gittings L, Odong Lukone S, Kisubi N, Atama M, Kyambadde P. Todurujo na Kadurok (empowering youth): study protocol of an HIV self-testing and edutainment comic cluster randomised trial among refugee youth in a humanitarian setting in Uganda. BMJ Open. 2022 Nov 23;12(11):e065452. doi: 10.1136/bmjopen-2022-065452. PMID 36418143